CLINICAL TRIAL: NCT03782883
Title: The Impact of Charcot-Marie-Tooth Disease in the Real World
Status: Completed | Type: Observational
Sponsor: Vitaccess Ltd (Industry)
Collaborators: ACMT-Rete per la malattia di Charcot-Marie-Tooth OdV (Unknown); Charcot-Marie-Tooth Association (Other); Charcot-Marie-Tooth UK (Unknown); CMT France (Unknown); Federación Española de Enfermedades Neuromusculares (Unknown); Hereditary Neuropathy Foundation (Other Government); Pharnext S.C.A. (Other)
Responsible Party: Principal Investigator, Mark Larkin, Director, Vitaccess Ltd
Other Study IDs: 5101-01-2018
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-04

CONDITIONS: Charcot-Marie-Tooth Disease
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 62 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
An observational, non-interventional registry study to collect real-world data from people living with Charcot-Marie-Tooth disease (CMT) and its treatment, which will be available to researchers to further the knowledge of Charcot-Marie-Tooth disease and improve patient care.

DETAILED DESCRIPTION:
The registry uses Vitaccess' digital real-world evidence platform and has been developed in collaboration with CMT experts, Patient Advocacy Organizations (PAOs) and the biopharmaceutical company Pharnext.

Eligible participants install a study app on their smartphone. Researchers access aggregated, anonymised data via a cloud-based research portal.

The platform provides benefits to participants, which it is hoped will encourage persistence with data submission; these include options to download a copy of their symptom diary, a clinically-validated Knowledge feature, and access to high-level results from the study data.

The aggregated data are available in close to real time via "dashboards" and can be analysed according to a number of pre-set criteria (e.g. disease stage, age, geographic location).

State-of-the-art technologies and security policies are used in the platform to ensure industry-standard data storage and privacy for all users. Participants' personally identifiable information will remain confidential at all times, and researchers will not be able to identify individuals.

The study is ethics-approved in all scope countries and led by a Scientific Advisory Board comprising representatives from international PAOs, patients and key opinion leaders from each country, and study leads from both Pharnext Société Anonyme (SA) and Vitaccess Ltd.

ELIGIBILITY:
Inclusion Criteria:

(*) Aged 18 years and over (*) Diagnosed with any stage and any subtype of Charcot-Marie-Tooth disease (*) Resident in France, Germany, Italy, Spain, the UK, or the USA (*) Have a National Health Service (NHS) or Community Health Index (CHI) number, or equivalent (*) Willing to use their own smartphone

Exclusion Criteria:

(*) No specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (age >18 years) with any stage and any subtype of Charcot-Marie-Tooth disease, who are resident in France, Germany, Italy, Spain, the United Kingdom (UK) or the USA, so long as they have a National Health Service (NHS) or Community Health Index (CHI) number (or equivalent) and are willing to use their own smartphone / tablet.
Sampling Method: Non-Probability Sample
Enrollment: 3321 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
EuroQoL 5-dimension 5-level (EQ-5D-5L) | Throughout study completion, up to 62 months
  The EQ-5D-5L comprises two parts - the EQ-5D-5L descriptive system and the EQ Visual Analogue Scale (EQ VAS).
  The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, and anxiety/depression), each with 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems - i.e., higher scores represent worse health). The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.
  The EQ VAS records the respondent's self-rated health on vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. Higher scores represent better self-perceived health.

SECONDARY OUTCOMES:
Work Limitations Questionnaire (WLQ) | Throughout study completion, up to 62 months
  The WLQ measures the impact of CMT on participants' work ability and productivity. The measure comprises 25 items that ask respondents to rate their level of difficulty or ability to perform specific job demands, aggregated into four domains: time management, physical demands, mental-interpersonal demands, and output demands. Domain scores range from 0 to 100 and the recall period is the previous 2 weeks. WLQ domain scores can be converted into an estimate of productivity loss using an algorithm.
Brief Fatigue Inventory (BFI) | Throughout study completion, up to 62 months
  The BFI assesses the fatigue severity in patients with CMT. The measure comprises 10 items, although the first item asks about usual fatigue over the past week (with the respondent answering "yes" or "no") and is not included in the overall score. The remaining nine items assess general fatigue within two subscales: fatigue severity (three items), and the impact of fatigue on daily functioning (six items). The measure uses a 10-point numeric rating scale, and a recall period of 24 hours. A global fatigue score can be calculated by averaging all nine items.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity 3a and Interference 8a | Throughout study completion, up to 62 months
  The PROMIS pain intensity measure includes two items that assess pain intensity over the last 7 days (average and worst pain), and one for pain intensity "right now"; each scores using a 5-point scale. Scores range from 2-10. Higher scores represent worst pain. This measure is generic rather than disease-specific.
  The PROMIS pain interference measure assesses the extent to which pain hinders engagement with social, cognitive, emotional, physical and recreational activities, sleep, and enjoyment in life over the last 7 days using a 5-point scale. Scores range from 8-40. Higher scores represent worse interference. This measure is generic rather than disease-specific.
Bespoke questionnaire for this study | Throughout study completion, up to 62 months
  Two cramp-specific items were developed for inclusion in the survey, measuring cramp frequency and intensity. The cramp frequency item asks "In the past 7 days, how many days did you experience cramp?" and has five possible responses: had no cramp, 1-2 days, 3-4 days, 5-6 days, every day. The cramp intensity item asks "In the past 7 days, how intense was your cramp at its worst?" and has five possible responses: had no cramp, mild, moderate, severe, very severe. Higher scores on both items represent greater cramp frequency and intensity respectively.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance 8a | Throughout study completion, up to 62 months
  The PROMIS sleep disturbance measure assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep over the last 7 days using a 5-point scale. Scores range from 8-40. Higher scores represent worse sleep disturbance. This measure is generic rather than disease-specific.
Falls Efficacy Scale - International (FES-I) | Throughout study completion, up to 62 months
  The FES-I measures the level of concern about falling during social and physical activities inside and outside hte home, whether or not the person actually does the activity. The "usual" level of concern is measured on a four-point Likert scale (1 = not at all concerned to 4 = very concerned), with a time frame of "usual". Scores range from 16-64. Higher scores represent greater concern about falling.
Lower Extremity Function Scale (LEFS) | Throughout study completion, up to 62 months
  The LEFS evaluates difficulties because of lower limb problems in 20 activities, including work/school activities, hobbies, moving around the home, dressing, lifting, standing, sitting, walking, and running. The level of difficulty is assessed for "today" using a 5-point Likert scale (0 = extreme difficulty or unable to perform activity; 5 = No difficulty). Lower scores represent greater difficulties experience because of lower limb problems.
QuickDash (Disabilities of the Arm, Shoulder and Hand) | Throughout study completion, up to 62 months
  The QuickDash measure uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. Six questions relate to the ability to perform six activities over the last week, ranging from opening a jar, carrying, washing and recreational activities; two questions relate to impact on social and daily activities; two questions ask the person to rate the severity of pain and tingling in the arms, shoulder or hand, and one question relates to the effects of pain on sleep. All questions are rated 1-5 (no difficulty/none/not at all through to unable/extreme difficulty). Scores range from 11-55. Higher scores represent greater difficulties with physical function and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mark JW Larkin, PhD, Principal Investigator — Vitaccess Ltd
Locations (1):
- Vitaccess Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Aggregated data research dashboards will be available via industry subscriptions or free academic access.

REFERENCES:
- [Background] Thomas FP, Saporta M, Attarian S, Sevilla T, Mascaro RS, Fabrizi GM, Genovese F, Gray A, Bull S, Tanesse D, Rego M, Moore A, Hollett C, Monteiro K, Paoli X, Llewellyn S, Larkin M, Boutalbi Y. Patient-reported impact of Charcot-Marie-Tooth disease: protocol for a real-world digital lifestyle study. Neurodegener Dis Manag. 2021 Feb;11(1):21-33. doi: 10.2217/nmt-2020-0044. Epub 2020 Oct 22. PMID 33086913
- [Background] Thomas FP, Saporta MA, Attarian S, Sevilla T, Sivera R, Fabrizi GM, Genovese F, Gray AJ, Bull S, Tanesse D, Rego M, Moore A, Hollett C, Paoli X, Senechal T, Day L, Ouyang C, Llewellyn S, Larkin M, Boutalbi Y. Patient-Reported Symptom Burden of Charcot-Marie-Tooth Disease Type 1A: Findings From an Observational Digital Lifestyle Study. J Clin Neuromuscul Dis. 2022 Sep 1;24(1):7-17. doi: 10.1097/CND.0000000000000426. Epub 2022 Aug 19. PMID 36005469
- See also: Research portal via which anonymised data can be made available to approved researchers — https://vitaccess.com/charcot-marie-tooth-disease-dataset/
- See also: Registration page to enrol in the study — https://vitaccess.com/cmt-and-me/
- See also: Digital platform used to support the study — https://vitaccess.com/